CLINICAL TRIAL: NCT03502603
Title: Pilot Study of New Computer-based Neuropsychological Tool: Visual Tests, Touch Responses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 17-01677
Record Dates: First submitted 2018-04-11; First posted 2018-04-18 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Cerebral Neurological Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cerebral neurological illness (CNI) participants (Active Comparator): Identified from the department of Rehabilitation, Psychiatry, and Medicine and referred to the research staff via in-person communication, email or staff message
  Interventions: Diagnostic Test: Railroad Test; Diagnostic Test: Swamp Test; Diagnostic Test: Presidents Recognition Test; Diagnostic Test: Judgment of Line Orientation; Diagnostic Test: Symbol Span subtest of the Wechsler Memory Scale-IV; Diagnostic Test: Information subtest of the Wechsler Adult Intelligence Scale-IV:; Diagnostic Test: Digit Span subtest of the Wechsler Adult Intelligence Scale-I; Diagnostic Test: Reading subtest of the Wide Range Achievement Test; Diagnostic Test: Symbol Digit Modalities Test:; Diagnostic Test: Dot Counting Test
- Non-CNI participants (Active Comparator): Identified from the department of Rehabilitation, Psychiatry, and Medicine and referred to the research staff via in-person communication, email or staff message
  Interventions: Diagnostic Test: Railroad Test; Diagnostic Test: Swamp Test; Diagnostic Test: Presidents Recognition Test; Diagnostic Test: Judgment of Line Orientation; Diagnostic Test: Symbol Span subtest of the Wechsler Memory Scale-IV; Diagnostic Test: Information subtest of the Wechsler Adult Intelligence Scale-IV:; Diagnostic Test: Digit Span subtest of the Wechsler Adult Intelligence Scale-I; Diagnostic Test: Reading subtest of the Wide Range Achievement Test; Diagnostic Test: Symbol Digit Modalities Test:; Diagnostic Test: Dot Counting Test

INTERVENTIONS:
Diagnostic Test: Railroad Test — This is a test designed to evaluate visual perception capacities and requires the participant to match photographs with railroads as a central theme. The participant is presented with a photograph image at the top of the screen and is asked to match it to one of the two, three or four choices in the lower portion of the display.
  Other Names: 1 Day
Diagnostic Test: Swamp Test — This is a test of immediate visual memory/attention for photographs with swamp wetlands as a central theme. The participant is briefly presented with a photograph which is replaced by two, three or four choices, one of which the participant is asked to select as the initially presented image.
Diagnostic Test: Presidents Recognition Test — This is a test of history knowledge and facial recognition using pictures of US presidents and non-president distractors. The participant is presented with two photographs and is asked to identify which is the picture of a US president
Diagnostic Test: Judgment of Line Orientation — This test requires participants to visually match the orientation of line segments. This is a test of visual perception and was included as a relative equivalent of the Railroad Test.
Diagnostic Test: Symbol Span subtest of the Wechsler Memory Scale-IV — This test requires participants to immediately recall a sequence of designs after a brief presentation. This is a test of immediate visual memory/attention and was included as a relative equivalent of the Swamp Test
Diagnostic Test: Information subtest of the Wechsler Adult Intelligence Scale-IV: — This test requires participants to answer factual knowledge questions. This is a test of fund of knowledge and was included as a verbal equivalent for the non-verbal Presidents Recognition Test.
Diagnostic Test: Digit Span subtest of the Wechsler Adult Intelligence Scale-I — This test requires the participant to repeat sets of digits forward, backward, and to sequence digits in ascending order. This is a test of immediate memory/attention and was included to investigate possible attentional correlates of the Swamp Test. This test includes a performance validity indicator that will permit analyses of validity indicators included with the experimental tests
Diagnostic Test: Reading subtest of the Wide Range Achievement Test — This test requires participants to read words printed on a card. This is a test of word knowledge/academic achievement and was included to investigate the academic achievement concomitants of the Presidents Recognition Test.
Diagnostic Test: Symbol Digit Modalities Test: — This test requires participants to visually match abstract symbols with numbers within a certain time period. The participant either verbalizes or writes the response on an answer sheet. This is a test of speed of information processing and was included to assess speed of response factors pertaining to all of the experimental tests as reflecting speed of information processing.
Diagnostic Test: Dot Counting Test — This test requires participants to count arrays of dots presented on a card while being timed. This is a performance validity test and was included to ascertain validity factors pertaining to each of the experimental tests.

SUMMARY:
This study is aimed at investigating three new tests that will form part of a computerized tool designed to test brain/cognitive functioning. The system will be evaluated along with the tests' usability on samples of healthy controls and neurologically impaired patient participants. These new tests will be assessed with regard to reliability and validity. Reliability will be addressed through investigation of internal consistency of the test items. Validity will be evaluated relative to traditional paper-and-pencil tests and differentiation between patient and healthy participants.Each participant will complete both the computerized and paper and pencil-based tests. The results will be analyzed to see how performances on the two test types compare. The overall aim of this project is to determine if these new computerized tasks are an improvement over standard paper and pencil-based neuropsychological measures.

ELIGIBILITY:
Inclusion Criteria:

Individuals without positive cerebral findings on neuroimaging (Non-PCF)

* Participants can be male or female and between the ages of 21 and 65 years old.
* Participants will have adequate perceptual and motor capabilities to participate in testing.

Neuroimaging-positive cerebral findings (PCF)

* Patients at NYULMC identified to have significant cerebral findings on neuroimaging.
* Participants will be male or female and between the ages of 21 and 65 years old.
* Participants will have adequate perceptual and motor capabilities to participate in testing.

Exclusion Criteria:

* Participants without adequate perceptual and motor capacities preventing them from participation in the testing.
* Participants with severe dysfunction at the level of dementia that can interfere with informed consent.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2019-05-10 (Actual); Primary Completion 2023-12-06 (Actual); Study Completion 2023-12-06 (Actual)

PRIMARY OUTCOMES:
Score on Railroad Test | 1 Day
Score on Swamp Test | 1 Day
Score on President Recognition Test | 1 Day

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Chervinsky, PhD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Requests should be directed to alexander.chervinsky@nyulangone.org . To gain access, data requestors will need to sign a data access agreement.